CLINICAL TRIAL: NCT02507154
Title: Phase I/II Study of Expanded, Activated Autologous Natural Killer Cell Infusions With Cetuximab for Patients With EGFR-Positive Nasopharyngeal Carcinoma or Head and Neck Squamous Cell Carcinoma
Brief Title: Reactivating NK Cells in Treating Refractory Head and Neck Cancer
Acronym: NKEXPHNC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NK0906
Record Dates: First submitted 2015-07-22; First posted 2015-07-23 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Nasopharyngeal Cancer; Head and Neck Squamous Cell Carcinoma
Keywords: cetuximab; NK cells; nasopharyngeal cancer; head and neck squamous cell cancer
MeSH Terms: conditions — Nasopharyngeal Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cetuximab + NK cells (Experimental): During cycle 1, patient will receive intravenous cetuximab and subcutaneous IL-2 on day 1, followed by NK cell infusion on day 2, with subcutaneous IL-2 for an additional 5 doses three times a week to support NK cell viability and expansion in vivo. Following NK cell infusion, cetuximab will be administered weekly for another 2 weeks. During cycle 2 and 3, one cycle of cetuximab monotherapy will be administered 3 weeks apart. Patients who demonstrate objective tumor response or stable disease after cycle 3 will receive a second infusion of NK cells along with cetuximab during cycle 4 therapy at the same dose and schedule as in cycle 1. This will be followed by 2 additional cycles of cetuximab monotherapy (3 weeks apart).
  Interventions: Drug: Cetuximab + NK cells

INTERVENTIONS:
Drug: Cetuximab + NK cells
  Other Names: Erbitux

SUMMARY:
This study aims to determine the safety and efficacy of expanded activated autologous NK cells administered after cetuximab in patients with EGFR-positive nasopharyngeal carcinoma or head and neck squamous cell carcinoma.

DETAILED DESCRIPTION:
Natural killer (NK) cells are cytotoxic lymphocytes of the innate immune system that are responsible for direct and indirect cytolytic killing of virally-transformed and/or cancer cells. Harnessing NK cells in cancer immunotherapy therefore, provides a direct cytotoxic effect on cancer cells which further stimulates further downstream adaptive anti-tumor immune responses against the cancer. In order to effect a more targeted killing of these tumor cells, using a monoclonal antibody (mAb) to direct these NK cells to the target site is feasible, provided a specific tumor antigen can be identified. In nasopharyngeal Carcinoma (NPC) and head and neck squamous cell carcinoma (HNSCC) where epidermal growth factor receptor (EGFR) is ubiquitously expressed, combining NK cell therapy with cetuximab (a chimeric mouse/human anti-EGFR monoclonal antibody) to direct these NK cells against these EGFR tumor targets is possible. In this study, we seek to enhance the antitumor activity of cetuximab to treat EGFR-positive head and neck cancers by combing infusion of activated expanded autologous NK cells with cetuximab. Patients selected for this trial are those with refractory NPC and HNSCC where no feasible therapeutic options are available. This is a lead-in phase I followed by a phase II study. The phase I study will enroll 9 patients and will test the feasibility and safety of this combination strategy and determine the tolerated dose of NK cell infusion (1x1^06/kg or 1x10^7/kg NK cells) in adult EGFR positive NPC and HNSCC patients. For the first 3 patients, each new patient will only be enrolled at least 3 weeks after treatment of the preceding patient to allow sufficient time to monitor toxicities. Initial phase of treatment consists of 7 weeks of cetuximab monotherapy. At week 8, clinical evaluation will be done to determine patients who are suitable to continue this study with NK cell therapy, based on the severity of toxicities encountered. Eligible patients will undergo apheresis (Day -10) to harvest NK cells. The collected NK cells will be expanded and activated in the laboratory. During cycle 1, cetuximab will be given on day 1 with subcutaneous IL-2 (three times per week for 2 weeks); followed by expanded NK cells on day 2. The purpose of IL-2 is to sustain activity of these NK cells in-vivo. Cetuximab will be administered weekly for additional 2 weeks following the NK cell infusion during cycle 1. For cycle 2 and 3, cetuximab monotherapy will be administered every 21 days. Clinical evaluation will be performed upon completion of cycle 3. Patients with stable disease or with partial response will be allowed to continue with a second NK infusion dose as per cycle 1, followed by additional 2 more cycles of cetuximab monotherapy (every 21 days).

.

ELIGIBILITY:
Inclusion Criteria

1. Age >21
2. Histologically confirmed diagnosis of EGFR-positive nasopharyngeal carcinoma or EGFR positive HNSCC (based on >80% immunohistochemistry of biopsy of recurrent tumor Ventana (Roche) clone 3C6
3. Recurrent cancer that is not surgically salvageable
4. Metastatic disease (after one course of palliative chemotherapy has been completed)
5. Presence of measurable tumor by RECIST 1.1 criteria
6. At least two weeks since receipt of any biological therapy, chemotherapy, and/or radiation
7. Adequate organ function
8. Haemoglobin ≥ 9g/dL ANC ≥ 1500/µL Platelet count ≥ 100,000/µL Creatinine clearance ≥60ml/minute Total bilirubin ≤ 1.5 x upper limit normal (ULN) AST ≤ 5 x upper limit normal ALT ≤ 2 x upper limit normal INR and PTT <1.5 x upper limit normal (ULN)
9. ECOG performance status of 0-2
10. Life expectancy of at least 60 days
11. Localized radiotherapy for palliative pain management is permissible
12. Written consent to participate on study
13. Physiological dose of steroid replacement is permissible

Exclusion Criteria

1. Treatment within the last 30 days with any investigational drug
2. Hypersensitivity to cetuximab or any excipients of the NK cell product
3. Concurrent administration of any other tumor therapy, including cytotoxic chemotherapy, hormonal therapy, and immunotherapy
4. Major surgery within 28 days of study drug administration
5. Radiotherapy to the target lesions during study or within 3 weeks prior to study treatment.
6. Autologous bone marrow transplant
7. Active infection that in the opinion of the investigator would compromise the patient's ability to tolerate therapy
8. Lactating or pregnant
9. Unwilling to use adequate barrier contraception measures during study period.
10. Second primary malignancy that is clinically detectable at the time of consideration for study enrolment
11. Receipt of immunosuppressives or steroids (=1mg/kg) during time period of 3 days prior to expanded NK cell infusion to 30 days after infusion (i.e. day -3 to day +30).
12. Symptomatic brain metastases
13. Electrocardiogram with clinically significant findings.
14. Serious concomitant disorders that would compromise the safety of the patient or compromise the patient's ability to complete the study, at the discretion of the investigator; serious cardiac illness or medical conditions including but not limited to:

    * Patients with dyspnea at rest.
    * History of documented congestive heart failure
    * High risk uncontrolled arrhythmias
    * Angina pectoris requiring a medicinal product
    * Clinically significant valvular disease
    * Poorly controlled hypertension

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2015-07 (Actual); Primary Completion 2019-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Safety as measured by clinical examination including hematology, renal and liver function tests, adverse events and any significant biochemical abnormalities or toxicities | 12- 18 weeks
  During cycle 1 (21 days) and for at least 21 days following a second NK cell infusion if administered, patients will be reviewed twice a week. Clinical examination including hematology, renal and liver function tests will be performed. Any adverse events (using NCI CTC grading) and concomitant medications notation will be recorded. Any significant biochemical abnormalities or toxicities will be monitored till resolution of these findings or 30 days after patient withdraws from this study, whichever occurs later.
  During cycles with cetuximab monotherapy, patients with be reviewed once every cycle (21 days).
Objective tumor response | Up to 24 months
  In this study, treatment response will be determined using RECIST 1.1 criteria, after two and four cycles of therapy. The endpoints of the study are objective tumor response including overall response rate (ORR), partial response (PR), duration of complete response (DCR) and duration of partial response (DPR). Complete response is defined by complete resolution of target lesion while partial response is defined by reduction of the target lesion by at least 20% from its baseline. Duration of tumor response will be censored at the date of the last follow-up visit for tumor responders who are still alive and who have not progressed.

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital, Singapore, Singapore

REFERENCES:
- [Derived] Lim CM, Liou A, Poon M, Koh LP, Tan LK, Loh KS, Petersson BF, Ting E, Campana D, Goh BC, Shimasaki N. Phase I study of expanded natural killer cells in combination with cetuximab for recurrent/metastatic nasopharyngeal carcinoma. Cancer Immunol Immunother. 2022 Sep;71(9):2277-2286. doi: 10.1007/s00262-022-03158-9. Epub 2022 Jan 30. PMID 35098345